CLINICAL TRIAL: NCT05609058
Title: The Influence of Treatment Position (Prone vs. Supine) on Whole Breast Irradiation for Chinese Breast Cancer Patients :Comparative Study
Brief Title: The Influence of Treatment Position (Prone vs. Supine) on Whole Breast Target
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, NING_LI, professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-2019
Record Dates: First submitted 2022-10-24; First posted 2022-11-08 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer; radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Breast cancer patients with T1-T2N0M0 stage who underwent radiation therapy after conserving surgery were enrolled. Supine and Prone scan sets were acquired during free breathing for all patients. Target volumes and organs at risk (OARs) including heart, ipsilateral lung and bilateral breast were contoured by the same radiation oncologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast cancer underwent scanning in the supine position (Experimental): Breast cancer patients with T1-2N0M0 stage who underwent radiation therapy after conserving surgery were enrolled. Supine scan sets were acquired during free breathing for all patients. Target volumes and organs at risk (OARs) including heart, ipsilateral lung and bilateral breast were contoured by the same radiation oncologist. The tumor bed (TB) was determined based on surgical clips. The Clinical target volume (CTV)consisted of the whole breast. The planning target volume (PTV) was CTV plus 0.5cm. The boost of PTV (PTVboost) was TB plus 0.5cm.
  Interventions: Device: dedicated treatment board with no degree

INTERVENTIONS:
Device: dedicated treatment board with no degree — the patients were placed in the prone position on a dedicated treatment board with no degree incline using an arm support (with both arms above the head). Te board contained an open aperture on one side to allow for the ipsilateral breast to hang freely away from the chest wall

SUMMARY:
Radiotherapy after breast conserving therapy plays an important role in early stage breast cancer patients. It not only results in a reduction in local and regional recurrence but also decrease the death rate effectively. For adjuvant radiotherapy, supine positioning is the most common approach and has multiple advantages. Due to deformability and softness of the breast, during simulation and treatment in supine position, the breast stretches over the chest wall, especially in patients with large and pendulous glands. Thus the organs at risk (OARs) received dose increased. The radiotherapeutic toxicity are unavoidable. Some present studies show that the prone positioning of patients can improve dose homogeneity and reduce the dose distribution in OARs in patients with large and pendulous glands. Chinese women have relatively small breasts, the advantages of those have not been established. Therefore, investigators compared the parameters between supine and prone positions for whole breast irradiation after conserving surgery.

DETAILED DESCRIPTION:
Objective To investigate the difference of target volumes and dosimetric parameters between supine and prone positions for whole breast irradiation after conserving surgery.

Methods Breast cancer patients with T1-2N0M0 stage who underwent radiation therapy after conserving surgery were enrolled. Supine and Prone scan sets were acquired during free breathing for all patients. Target volumes and organs at risk (OARs) including heart, ipsilateral lung and bilateral breast were contoured by the same radiation oncologist. The tumor bed (TB) was determined based on surgical clips. The Clinical target volume (CTV)consisted of the whole breast. The planning target volume (PTV) was CTV plus 0.5cm. The boost of PTV (PTVboost) was TB plus 0.5cm. Dosimetric parameters of target volumes and OARs were compared between supine and prone position.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer patients with T1-T2N0M0 stage who underwent radiation therapy after conserving surgery
2. exhibited normal arm movement aſter surgery
3. had no chronic lung diseases
4. Written informed consent forms

Exclusion Criteria:

1. Breast cancer patients with radical surgery
2. could not exhibit normal arm movement after surgery
3. had chronic lung diseases
4. refused informed consent forms

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
dose distribution of GTV | 1 year
  the difference of GTV (Gross tumor target) between two plans
dose distribution of CTV | 1 year
  the difference of CTV (clinical target volume) between two plans
dose distribution of PTV | 1 year
  the difference of PTV (planing target volume) between two plans
dose distribution of heart | 1 year
  the difference of heart dose distribution between two plans
dose distribution of ipsilateral lung | 1 year
  the difference of ipsilateral lung dose distribution between two plans
dose distribution of bilateral breasts | 1 year
  the difference of bilateral breasts dose distribution between two plans

CONTACTS AND LOCATIONS:
Locations (1):
- Shanxi provicial cancer hospital, Taiyuan, Shanxi, China

REFERENCES:
- [Derived] Ma L, Yang Y, Ma J, Mao L, Li X, Feng L, Abulimiti M, Xiang X, Fu F, Tan Y, Zhang W, Li YX, Jin J, Li N. Correlation between AI-based CT organ features and normal lung dose in adjuvant radiotherapy following breast-conserving surgery: a multicenter prospective study. BMC Cancer. 2023 Nov 9;23(1):1085. doi: 10.1186/s12885-023-11554-2. PMID 37946125